CLINICAL TRIAL: NCT02545608
Title: A Randomised, Multi-centre, Evaluator-blinded, Split-hand, no Treatment-controlled Study to Evaluate the Safety and Efficacy of Restylane Vital for Skin Rejuvenation of the Dorsal Hands in Chinese Subjects
Brief Title: Safety and Efficacy of Restylane Vital for Skin Rejuvenation of Dorsal Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH1406
Record Dates: First submitted 2015-08-21; First posted 2015-09-10 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-06

CONDITIONS: Dorsal Hands

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Vital in both hands (Experimental): Open group used to develop a proper use of injection technique for Restylane Vital
  Interventions: Device: Restylane Vital
- Restylane Vital and No treatment (Other): Split-hand design: Restylane Vital in one hand and initially no treatment in the other hand
  Interventions: Device: Restylane Vital

INTERVENTIONS:
Device: Restylane Vital

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using Restylane Vital for skin rejuvenation of the dorsal hands. Assessment of improvement of skin structure will be done by a blinded evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Chinese origin
* Subject willing and able to comply with the requirements of the study and agrees to adhere to the visit schedule and to be compliant to the study instructions

Exclusion Criteria:

* Any previous non-permanent implant/filler in the hands
* Any mesotherapy or resurfacing procedure in the hands within 6 months prior to baseline
* Any previous hand surgery
* Any fibrosis or scarring or deformities on the hands
* Advanced photoaged/photodamaged skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (2):
- China (2):
  - Beijing
  - Shanghai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Vital in Both Hands | Restylane Vital in Randomized Hand, no Treatment in the Other
Started | 9 | 100 (Split hand study design. Total no. of subjects in Randomised group and No-treatment control is 100.)
Completed | 9 | 93
Not Completed | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Vital in Both Hands | Restylane Vital in Randomized Hand, no Treatment in the Other | Total
Number analyzed (Participants) | 9 | 100 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 92 | 101
  >=65 years | 0 | 8 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (8.2) | 48.5 (11.2) | 48 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 96 | 105
  Male | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  China | 9 | 100 | 109

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of Restylane Vital on Skin Structure Compared to no Treatment Using a Validated Scale.
Description: Assessment of the severity of hand aging using a 5-point (ranging from 0-5) photo numeric rating scale (Hand Grading Scale), where higher scores mean a worse outcome.
Time Frame: 12 weeks
Population: The 9 subjects treated with Restylane Vital in both hands not included
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Restylane Vital in Randomized Hand: Restylane Vital in randomized hand
- No-treatment Control Hand: No treatment control hand
Arm/Group | Restylane Vital in Randomized Hand | No-treatment Control Hand
Number analyzed (Participants) | 100 | 100
units on a scale | 0.85 (0.59) | 2.17 (0.49)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months (AE reporting on each subject started at visit 2 and continued during each follow-up visit (including telephone contacts and extra visits between planned visits) until the last scheduled visit in the study.)
Description: Each subject should be questioned about AEs at each study visit following the screening visit.
  The question asked should be:"Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from signs and symptoms detected during each examination, observations made by the study site personnel, subject diaries, or spontaneous reports from the subjects.
Groups:
- Restylane Vital in Both Hands: Restylane Vital in both hands
Arm/Group | Restylane Vital in Both Hands | Restylane Vital in Randomized Hand | No-treatment Control Hand
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/100 | 2/100
Other Adverse Events (participants affected / at risk) | 0/9 | 12/100 | 3/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Vital in Both Hands (N=9) | Restylane Vital in Randomized Hand (N=100) | No-treatment Control Hand (N=100)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Worsening of lumbar disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Vital in Both Hands (N=9) | Restylane Vital in Randomized Hand (N=100) | No-treatment Control Hand (N=100)
Implant site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 4 (4) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 4 (4) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 4 (4) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other